CLINICAL TRIAL: NCT02860897
Title: Patient Adherence to Premarin Versus Vagifem Therapy After Female Pelvic Reconstructive Surgery
Status: Withdrawn | Phase: Phase 4 | Type: Interventional
Why Stopped: Unable to provide study medications due to cost.
Sponsor: University Hospitals Cleveland Medical Center (Other)
Responsible Party: Principal Investigator, Andrey Petrikovets, Fellow in Female Pelvic Medicine and Reconstructive Surgery, University Hospitals Cleveland Medical Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 08-15-39
Record Dates: First submitted 2016-07-28; First posted 2016-08-09 (Estimated); Last update posted 2018-05-02 (Actual); Status verified 2018-04

CONDITIONS: Estrogen; Menopause; Pelvic Floor Disorders; Surgery
MeSH Terms: conditions — Pelvic Floor Disorders | interventions — Estrogens, Conjugated (USP); Estradiol

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Vaginal estrogen cream (Experimental)
  Interventions: Drug: Premarin
- Vaginal estrogen tablet (Experimental)
  Interventions: Drug: Vagifem

INTERVENTIONS:
Drug: Premarin — Vaginal estrogen cream
  Arms: Vaginal estrogen cream
Drug: Vagifem — Vaginal estrogen tablet
  Arms: Vaginal estrogen tablet

SUMMARY:
PURPOSE: To evaluate patient adherence to cream versus tablet based local estrogen therapy by randomizing treatment modalities to determine differences in adherence to either form.

HYPOTHESIS: There is no difference in adherence to cream versus tablet based local estrogen therapy when prescribed as a 6 week course of postoperative therapy after female pelvic reconstructive surgery.

DETAILED DESCRIPTION:
Genitourinary syndrome is the consequence of the lack of estrogen exposure to the genitourinary tract during menopause. The result of this hypoestrogenic state is the thinning, shrinking, increased vaginal friction, and increase in lower urinary tract symptoms. It is estimated that up to 60% of postmenopausal women experience these symptoms and the widely accepted treatment for genitourinary syndrome is the application of local estrogen.

Estrogen has been widely prescribed as a beneficial adjunct in the treatment of menopausal genitourinary syndrome and is used to decrease the incidence of urgency, frequency, nocturia, stress urinary incontinence, urge urinary incontinence, and recurrent urinary tract infections. Despite the well described use of local estrogen therapy for genitourinary syndrome, not all forms of vaginal estrogen are created equally and patient adherence to prescriptions has not been uniform among different formulations. Shulman and colleagues noted that when used for genitourinary syndrome, patients who were prescribed local estrogen tablets demonstrated significantly longer compliance to therapy than those prescribed estrogen cream (149 days vs. 92 days). Similarly, in a cohort of 30,000 patients, Portman demonstrated that patients prescribed vaginal estrogen tablets were also more likely to be adherent to therapy than those given the cream formulation. Some of the reasons for early discontinuation of local vaginal cream was due to messiness with application, leakage, concerns about underdosing or overdosing, and that the cream was generally unpleasant.

Given the extensive use of local estrogen for genitourinary syndrome, despite limited data, surgeons have been prescribing local estrogen to prevent the development of postoperative complications like lower urinary tract symptoms after female pelvic reconstructive surgery. In a postoperative 12 week follow up, Karp and colleagues noted that the administration of a vaginal estrogen tablets in postmenopausal women is associated with improved vaginal maturation indices and objective atrophy assessment after vaginal reconstructive surgery. Vaccaro also noted that preoperative administration of vaginal estrogen administered 2- 12 weeks before reconstructive surgery improves the vaginal maturation index by more than 15.5% and may improve the tissue as a substrate for suture placement. There have been two studies evaluating the effect of vaginal estrogen after midureteral sling placement: Zullo studied retropubic midureteral slings and noted that patients who did not receive vaginal estrogen tablets exhibited a higher incidence of urinary urgency than patients who did (4% vs. 29%). Liapias evaluated local estrogen application for 6 months after transobturator tape slings and noted statistically significant decreases in urinary frequently and urgency.

Given this data, there appears to be a role for postoperative local estrogen therapy after pelvic reconstructive surgery but it not clear if patients are adherent to therapy and the form of therapy: cream or tablet. To the best of the investigators knowledge, there is no data that describes patient adherence to local estrogen therapy after female pelvic surgery. Therefore, the purpose of this study is to evaluate patient adherence to cream versus tablet based local estrogen therapy by randomizing treatment modalities to determine differences in adherence to either form.

ELIGIBILITY:
Inclusion Criteria:

* Patients who underwent female pelvic reconstructive surgery at University Hospitals Case Medical Center and were given postoperative local estrogen therapy.
* Patients who consented to the study.
* Postmenopausal

Exclusion Criteria:

* Patients who were not given a prescription for postoperative lower estrogen therapy despite undergoing surgery.
* Patients with contraindications to vaginal estrogen.
* Any obliterative procedures. Patients who are unable to participate in informed consent. Patients younger than 18. Non English speaking patients

Ages: 18 Years to 90 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2016-07; Primary Completion 2017-04 (Estimated); Study Completion 2017-07 (Estimated)

PRIMARY OUTCOMES:
Time in days to discontinuation of vagifem tablet or premarin cream. | 6 weeks
  Days upon which patients stopped using vagifem tablets or premarin cream

SECONDARY OUTCOMES:
Pelvic floor disease inventory-20 | preoperatively, 2 weeks, 6 weeks.
  The investigators will use the pelvic floor disease inventory-20 survey and compare its results preoperatively, 2 weeks and 6 weeks after surgery.
Postoperative complications | 6 weeks

CONTACTS AND LOCATIONS:
Locations (1):
- University Hospitals Case Medical Center, Cleveland, Ohio, United States

IPD SHARING:
Plan to Share IPD: No